CLINICAL TRIAL: NCT04778189
Title: Effect of Intravenous Dexamethasone on the Duration of Hyperbaric Bupivacaine Spinal Anesthesia in Lower Abdominal Surgery, Randomized Controlled Trial
Brief Title: Effect of Intravenous Dexamethasone on Duration of Hyperbaric Bupivacaine Spinal Anesthesia in Lower Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AssiutU_dexamethasone
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Spinal Anesthesia
Keywords: i.v dexamethasone; hyperparic bupivacaine

STUDY DESIGN:
Intervention Model Description: patients will be scheduled for lower abdominal surgery under spinal anesthesia will randomly be allocated into two groups, group SD and group SN, After placement of standard monitors and peripheral IV access, with aseptic technique we will insert, a 25-G pencil-point Pencan(B. Braun, Mississauga, Ontario, Canada) needle intrathecally at the L4-5 or L3-4 interspace, with the patient in a seated position. We will confirm Intrathecal positioning by observation of cerebrospinal fluid return through the needle. Then we will inject the hyperbaric bupivacaine. All patients will receive spinal anesthesia with 12-mg hyperbaric bupivacaine 0.5%. Patients will be randomly assigned to one of the 2 Groups. Beginning during the intrathecal injection, patients in group( SD )will receive 8-mg dexamethasone IV in 500-mL normal saline (total, 502 mL), while patients in group( NS ) will receive 500-mL normal saline IV in 5-10 minutes,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline group (NS) (Placebo Comparator): patients in group( NS ) will receive 500-mL normal saline IV in 5-10 minutes after spinal anesthesia
  Interventions: Drug: Placebo
- dexamethasone group (SD) (Active Comparator): patients in group( SD )will receive 8-mg dexamethasone IV in 500-mL normal saline in 5-10 minutes after spinal anesthesia
  Interventions: Drug: i.v dexmethasone

INTERVENTIONS:
Drug: Placebo — while patients in group( NS ) will receive 500-mL normal saline IV in 5-10 minutes, after spinal anesthesia
  Arms: normal saline group (NS)
Drug: i.v dexmethasone — patients in group( SD )will receive 8-mg dexamethasone IV in 500-mL normal saline after spinal anesthesia
  Arms: dexamethasone group (SD)

SUMMARY:
The use of dexamethasone, administered either systemically or perineurally, as an adjunct to peripheral or neuraxial regional blocks, is currently one of the hottest topics in the field of regional anesthesia.

DETAILED DESCRIPTION:
A large number of clinical studies have investigated this off-label application of dexamethasone in recent years, with many reporting enhanced sensory block and/or improved postoperative analgesia following either intravenous (i.v.) or perineural dexamethasone. Dexamethasone is potent, selective glucocorticoid having minimal mineralocorticoid action. Systemic anti-inflammatory and immunosuppressive properties may be responsible for the prolongation of analgesia when administered intravenously. Various studies proved the efficacy of steroids for the prolongation of the effects of regional nerve blocks. We decided to conduct the present study to evaluate the effects of intravenous (IV) dexamethasone on the subarachnoid block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists score I-III,
* Patients undergoing lower abdominal surgery under hyperbaric bupivacaine spinal anesthesia

Exclusion Criteria:

* History of allergy to amide LAs or dexamethasone,
* Presence of a preexisting lower limb neurological deficit
* Chronic use of corticosteroids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
regression of sensory block | 5, 10, 20, and 30 minutes after injection of local anesthetic(LA)
  Onset to regression of 2 dermatomes evaluated using a Von Frey6.1-g filament (Bioseb; North Coast Medical, Gilroy, CA)

CONTACTS AND LOCATIONS:
Overall Officials: Amani H Abdel-wahab, MD, Principal Investigator — Assiut University
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Wahab AH, Abd Alla ES, Abd El-Azeem T. Effect of intravenous dexamethasone on the duration of hyperbaric bupivacaine spinal anesthesia in lower abdominal surgery, Randomized controlled trial. BMC Anesthesiol. 2023 Sep 22;23(1):323. doi: 10.1186/s12871-023-02282-y. PMID 37736711